CLINICAL TRIAL: NCT00967824
Title: Developing and Testing a Tamoxifen Prophylaxis Decision Aid
Brief Title: Tamoxifen Citrate Decision Aids for Women at Increased Risk of Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Peter Anthony Ubel, University of Michigan Comprehensive Cancer Center
Allocation: Randomized
Other Study IDs: CDR0000649906; P50CA101451 (NIH); P30CA046592 (NIH); IRBMED-2004-0695 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Other: informational intervention
Other: questionnaire administration
Other: survey administration

SUMMARY:
RATIONALE: Evaluating a decision aid that describes the risks and benefits of taking tamoxifen citrate to prevent breast cancer may be helpful for women at increased risk of breast cancer.

PURPOSE: This randomized phase I/II trial is studying tamoxifen citrate decision aids for women at increased risk of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop and test a decision aid for describing the risks and benefits of taking tamoxifen citrate to prevent primary breast cancer in women at increased risk of breast cancer.

OUTLINE:

* Phase I: Patients are randomized to view 1 of 16 decision aids that vary in terms of how the information is presented based on 5 dimensions: 1) statistical information in pictographs vs plain text, 2) risk information presented with denominators of 100 vs 1000, 3) risk information presented in terms of total vs additional risk, 4) whether the risks of tamoxifen citrate are presented before or after the benefits are presented, and 5) contextual information about other risks the patient faces (all cause mortality, colon cancer, heart attack).

Patients complete baseline and post-test questionnaires.

* Phase II: Patients are randomized to 1 of 3 arms.

  * Arm I (control): Patients do not view the decision aid, but complete baseline and post-test questionnaires.
  * Arm II (control): Patients complete a baseline questionnaire only. They do not view the decision aid or complete the post-test questionnaire.
  * Arm III (intervention): Patients view 1 of 16 decision aids that vary based on 5 factors: 1) providing (or not) comparative information about the average woman's breast cancer risk, 2) sequencing presentation of risks and benefits (risks first vs benefits first), 3) including (or not) a summary table following presentation of risks and benefits, 4) using second vs third person language ("your risk" vs "a person like you"), and 5) presenting the decision as having 2 vs 3 options (taking/not taking a breast cancer prevention drug vs taking tamoxifen citrate/raloxifene, or no drug). Patients also complete baseline and post-test questionnaires.

Patients in both phases complete an online follow-up survey at 3 months. Patients in arms I or II (of phase II) receive a decision aid after completion of the follow-up survey.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Believed to be at increased risk of breast cancer (risk of ≥ 1.66% over 5 years) according to electronic-based medical data

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1683 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Development and testing of a decision aid that describes the risks and benefits of taking tamoxifen citrate to prevent primary breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fagerlin, PhD, Principal Investigator — University of Michigan Rogel Cancer Center

REFERENCES:
- [Derived] Korfage IJ, Fuhrel-Forbis A, Ubel PA, Zikmund-Fisher BJ, Greene SM, McClure JB, Smith DM, Alford SH, Fagerlin A. Informed choice about breast cancer prevention: randomized controlled trial of an online decision aid intervention. Breast Cancer Res. 2013;15(5):R74. doi: 10.1186/bcr3468. PMID 24004815
- [Derived] Banegas MP, McClure JB, Barlow WE, Ubel PA, Smith DM, Zikmund-Fisher BJ, Greene SM, Fagerlin A. Results from a randomized trial of a web-based, tailored decision aid for women at high risk for breast cancer. Patient Educ Couns. 2013 Jun;91(3):364-71. doi: 10.1016/j.pec.2012.12.014. Epub 2013 Feb 8. PMID 23395006